CLINICAL TRIAL: NCT01220570
Title: A Clinical Trial to Qualify the Growth Factor Signature (GFS) as an Intermediate Biomarker of Response for Development of PI3K-Pathway Inhibitors in Patients With Breast Cancer
Brief Title: The Growth Factor Signature (GFS) as an Intermediate Biomarker of Response for Development of PI3K-Pathway Inhibitors in Patients With Breast Cancer (MK-8669-050)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-050
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; ridaforolimus; ridaforolimus/dalotuzumab combination therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ridaforolimus; dalotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ridaforolimus + Dalotuzumab (Experimental): Ridaforolimus (MK-8669) + Dalotuzumab (MK-0646)
  Interventions: Drug: Ridaforolimus + Dalotuzumab
- Ridaforolimus (Experimental): Ridaforolimus (MK-8669)
  Interventions: Drug: Ridaforolimus
- Dalotuzumab (Experimental): Dalotuzumab (MK-0646)
  Interventions: Drug: Dalotuzumab

INTERVENTIONS:
Drug: Ridaforolimus + Dalotuzumab — Ridaforolimus (MK-8669) once daily for 5 consecutive days per week and Dalotuzumab (MK-0646) intravenously (IV) once weekly for 2 weeks
  Other Names: MK-8669, MK-0646
  Arms: Ridaforolimus + Dalotuzumab
Drug: Ridaforolimus — Ridaforolimus 40 mg (once daily for 5 consecutive days per week) for 2 weeks, 10 mg enteric-coated tablets
  Other Names: MK-8669
  Arms: Ridaforolimus
Drug: Dalotuzumab — Dalotuzumab, intravenously (IV) at 10 mg/kg/week for 2 weeks
  Other Names: MK-0646
  Arms: Dalotuzumab

SUMMARY:
This clinical trial will evaluate whether treatment with ridaforolimus, dalotuzumab, or ridforolimus/dalotuzumab combination therapy reduces Growth Factor Signature (GFS) Score among participants with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant has operable Stage I-IIIa invasive breast cancer of the following subtype: ER-positive, HER2-negative tumor with histologic grade 2 or 3 and Ki67 ≥ 15%
* Tumor is at least 2 cm in diameter as assessed by physical or radiographic exam
* Participant consents to provide an existing tissue sample or to have a core needle biopsy before drug administration
* Participant consents to provide tissue samples following drug administration by a second core needle biopsy or from a surgical specimen
* Participant must have adequate organ function

Exclusion Criteria:

* Participant has received any prior chemotherapy, biological therapy or radiotherapy for breast cancer
* Participant has a known hypersensitivity to the components of study drugs or their analogs, including hypersensitivity to macrolide antibiotics (e.g. clarithromycin, erythromycin, azithromycin).
* Participant has poorly controlled diabetes mellitus, or requires insulin for glucose control.
* Participant is unable to swallow capsules and/or absorb oral medications
* Participant is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study.
* Participant is known to be Human Immunodeficiency Virus (HIV)-positive
* Participant has known history of active Hepatitis B or C.
* Participant is concurrently using growth hormone (GH) or growth hormone inhibitors
* Participant has significant or uncontrolled cardiovascular disease, including heart failure, unstable angina, or a myocardial infarction within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The population mean change from baseline in GFS (Growth Factor Signature) score | Baseline and Day 15

SECONDARY OUTCOMES:
The population mean change from baseline in Ki67 among participants receiving ridaforolimus/dalotuzumab combination therapy | Baseline and Day 15
The correlation between change in Ki67 expression and change in GFS after two weeks of treatment with ridaforolimus/dalotuzumab (MK-8669/MK-0646) combination therapy, ridaforolimus (MK-8669) monotherapy and/or dalotuzumab (MK-0646) monotherapy | Baseline and Day 15